CLINICAL TRIAL: NCT01674153
Title: A Multi Protocol Investigation to Compare the Effects of Intra-dialytic Exercise on Physiological Changes and Toxin Removal in Maintenance Hemodialysis Patients
Brief Title: Investigating the Effects of Exercise on Physiological Changes and Toxin Removal in Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DSRB - 2011/01942; NKFRC/2011/01/06 (Other Grant/Funding Number: NKFRC/2011/01/06)
Record Dates: First submitted 2012-08-23; First posted 2012-08-28 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Renal Dialysis
Keywords: Intra-dialytic exercise; Toxin removal; Hemodiafiltration; Inter-compartmental resistance; Cardiac output

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HD-Exercise-HDF (Experimental): Prescribe intra-dialytic exercise of three bouts in 4 hours dialysis session.
  Interventions: Procedure: Intra-dialytic exercise

INTERVENTIONS:
Procedure: Intra-dialytic exercise — Perform intra-dialytic exercise of three bouts in 4 hours dialysis session. Each patient will perform exercise on Monark 881E rehab trainer (widely used in routine dialysis settings). The exercise intensity will be prescribed based on achievement of 50% of maximum heart rate for each recruited subject.

SUMMARY:
Hemodialysis is a life-saving treatment for end stage renal disease patients. The chief aims of hemodialysis are solute and fluid removal. Solute removal is associated with outcome of dialysis patients. Intra-dialytic exercise has been found to improve the toxin removal and it is suggested that exercise increases the cardiac output, thus increases the blood flow to lower extremities. This leads to increased toxin removal from low blood flow regions. On the other hand, exercise can possibly dilate the vasculature and decrease the compartmental resistance. In this study, the investigators aim to investigate the exercise induced physiological changes which enhances the toxin removal. This information combined with patient specific mathematical models will encourage clinicians to opt for Optimal intra-dialytic exercise protocol. On the other hand, Hemodiafiltration is widely accepted renal replacement therapy for improved toxin removal. Hence, we intend to compare the toxin removal outcome for standalone Hemodiafiltration and intra-dialytic exercise in conventional hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients male or female (Age > 21 years)
* Minimum dialysis vintage of 6 months
* Stable on hemodialysis
* Minimum Hemoglobin level of 10 g/dL
* Blood access capable of delivering the blood flow rate greater than 250 mL/min
* Preserved left ventricular ejection fraction (>50%) on prior imaging study
* Able to complete a 6min-walk-test without abnormal physiological response, excessive fatigue, or musculoskeletal discomfort

Exclusion Criteria:

* History of recurring or persistent hypotension in past 3 months
* Pregnant woman
* Severely Hypertensive patients (SBP > 180 mmHg and/or DBP > 115 mmHg)
* History of recent myocardial infarction or unstable angina (within past 6 months)
* Significant valvular disease, i.e. severe aortic stenosis and moderate-severe mitral regurgitation.
* Patients with end stage organ disease e.g. COPD, recent or debilitating CVA
* Patient with recent stroke (within past 6 months)
* Anemic patients
* History of known arrhythmia
* Participation in another clinical intervention trial
* Moderate to severe osteoarthritis of knee(s)
* Unable to consent

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-04 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Quantify toxin removal | 6 months
  Measure/estimate amount of toxin(s) removed and quantify corresponding physiological changes

SECONDARY OUTCOMES:
Compare exercise regimen with HDF | 6 months
  Compare amount of toxin removed for conventional hemodialysis (HD), HD with intra-dialytic exercise, and hemodiafiltration

CONTACTS AND LOCATIONS:
Overall Officials: Titus Lau, MD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- Dialysis Center, National University of Singapore, Singapore, Singapore

REFERENCES:
- [Background] Vaithilingam I, Polkinghorne KR, Atkins RC, Kerr PG. Time and exercise improve phosphate removal in hemodialysis patients. Am J Kidney Dis. 2004 Jan;43(1):85-9. doi: 10.1053/j.ajkd.2003.09.016. PMID 14712431
- [Result] Ward RA, Greene T, Hartmann B, Samtleben W. Resistance to intercompartmental mass transfer limits beta2-microglobulin removal by post-dilution hemodiafiltration. Kidney Int. 2006 Apr;69(8):1431-7. doi: 10.1038/sj.ki.5000048. PMID 16395268
- [Result] Maheshwari V, Samavedham L, Rangaiah GP. A regional blood flow model for beta2-microglobulin kinetics and for simulating intra-dialytic exercise effect. Ann Biomed Eng. 2011 Dec;39(12):2879-90. doi: 10.1007/s10439-011-0383-5. Epub 2011 Aug 30. PMID 21877220
- [Result] Parsons TL, Toffelmire EB, King-VanVlack CE. Exercise training during hemodialysis improves dialysis efficacy and physical performance. Arch Phys Med Rehabil. 2006 May;87(5):680-7. doi: 10.1016/j.apmr.2005.12.044. PMID 16635631
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639
- [Derived] Maheshwari V, Samavedham L, Rangaiah GP, Loy Y, Ling LH, Sethi S, Leong TL. Comparison of toxin removal outcomes in online hemodiafiltration and intra-dialytic exercise in high-flux hemodialysis: a prospective randomized open-label clinical study protocol. BMC Nephrol. 2012 Nov 23;13:156. doi: 10.1186/1471-2369-13-156. PMID 23176731